CLINICAL TRIAL: NCT05819866
Title: A Clinical Study to Assess the Efficacy and Safety of Leriglitazone in Adult Male Subjects With Cerebral Adrenoleukodystrophy
Acronym: CALYX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Minoryx Therapeutics, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-3-01
Record Dates: First submitted 2023-03-23; First posted 2023-04-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Adrenoleukodystrophy (cALD)
MeSH Terms: interventions — leriglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Leriglitazone (Active Comparator): Leriglitazone Treatment
  Interventions: Drug: Leriglitazone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leriglitazone — Leriglitazone at a strength of 15 mg/ml. Once-daily dosing at an initial volume of 10 ml
  Arms: Leriglitazone
Drug: Placebo — Placebo will match the study drug visually and by taste
  Arms: Placebo

SUMMARY:
A Clinical Study to Assess the Efficacy and Safety of Leriglitazone in Adults Male Subjects with Cerebral Adrenoleukodystrophy.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is male and aged ≥18 years.
* Subject has progressive cALD, defined as GdE+ brain lesions.
* Subjects for whom HSCT is not recommended by the investigator or subject is not willing to undergo HSCT.
* Subject has a Loes score ≥0.5 and ≤12 at Screening.
* Subject does not have major functional disability in the Major Functional Disabilities-Neurological Function Score (MFD-NFS), except for "wheelchair bound" or "total incontinence", which will be allowed as these are considered expected symptoms of AMN in the time course of the disease
* Subject does not have major cognitive impairment which would impair his ability to take part in the study as determined by the investigator at screening.

Key Exclusion Criteria:

* Subject who had previous bone marrow transplantation (HSCT) or treatment with ex-vivo gene therapy (eli-Cel).
* Subject has known type 1 or type 2 diabetes.
* Subject has known hypersensitivity or intolerance to pioglitazone or any other thiazolidinedione.
* Subject is taking or has taken honokiol, pioglitazone, or other thiazolidinediones within 3 months prior to Screening.
* Subject with current participation in another interventional clinical study or within 1 month prior to Screening.
* Subject with other medical, neuropsychiatric or social conditions that, in the opinion of the investigator, are likely to adversely affect the risk-benefit of study participation, interfere with study compliance, or confound the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the time to death or the subject becoming bedridden with a requirement for permanent ventilatory support, wichever comes earlier, in subjects treated with leriglitazone compared to placebo. | Interim analysis 1 (at 18 months of treatment)
  The primary endpoint will be the time to death or the subject becoming bedridden with a requirement for permanent ventilatory support, wichever comes earlier, in subjects treated with leriglitazone compared to placebo.
The primary endpoint will be the time to death or the subject becoming bedridden with a requirement for permanent ventilatory support, wichever comes earlier, in subjects treated with leriglitazone compared to placebo. | Interim analysis 2 (at 27 months of treatment)
  The primary endpoint will be the time to death or the subject becoming bedridden with a requirement for permanent ventilatory support, wichever comes earlier, in subjects treated with leriglitazone compared to placebo.
The primary endpoint will be the time to death or the subject becoming bedridden with a requirement for permanent ventilatory support, wichever comes earlier, in subjects treated with leriglitazone compared to placebo. | Final analysis (at 36 months of treatment)
  The primary endpoint will be the time to death or the subject becoming bedridden with a requirement for permanent ventilatory support, wichever comes earlier, in subjects treated with leriglitazone compared to placebo.

SECONDARY OUTCOMES:
Change from Baseline in Loes Score. | Interim analysis 1 (at 18 months of treatment)
  Change from Baseline in Loes Score. Loes Score Minimum = 0 Maximum =34 0 better outcome (healthy) 34 worst osutcome
Change from Baseline in Loes Score | Interim analysis 2 (at 27 months of treatment)
  Change from Baseline in Loes Score. Loes Score Minimum = 0 Maximum =34 0 better outcome (healthy) 34 worst osutcome
Change from Baseline in Loes Score | Final analysis (at 36 months of treatment)
  Change from Baseline in Loes Score. Loes Score Minimum = 0 Maximum =34 0 better outcome (healthy) 34 worst osutcome

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - Stanford University Medical Center, Palo Alto, California
  - Neuro Medicine Hospital / UF Health, Gainesville, Florida
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneota, Minnesota
  - Health University of Utah, Salt Lake City, Utah
- Hospital Austral, Buenos Aires, Argentina
- Federal University of Sao Paulo, São Paulo, Brazil
- ICM La Pitie Salpetriere, Paris, France
- Klinik und Poliklinik für Neurologie-Leipzig, Leipzig, Germany
- Sir Ganga Ram Hospital, New Delhi, India
- Hospital 12 de Octubre, Madrid, Spain
- National Hospital for Neurology and Neurosurgery, London, United Kingdom